CLINICAL TRIAL: NCT01693666
Title: Lifestyle Intervention Forever: Healthy Weight for Pregnancy and Birth (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Rosemary Catanzaro, RD, Registered Dietician, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22009; 8485 (Other: SLU eRS); 22009 (Other: SLU IRB)
Record Dates: First submitted 2012-09-10; First posted 2012-09-26 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy; Obesity; Weight Gain; Obstetric Complications
Keywords: Pregnancy; Obesity; Weight gain; Obstetric complications; Lifestyle intervention
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention group (Experimental): The LIFE program emphasizes improved nutritional quality, moderate physical activity, and weight maintenance (±10 lb) in obese pregnant women using a contingency management (CM) approach to reinforce behavior change. Participants will meet with the study dietitian and exercise physiologist every 2-4 weeks to develop and maintain individualized nutrition and physical activity plans, reinforced by CM. When the subject meets with the interventionists at their regular appointments, they will review the diet and exercise requirements, and provide vouchers earned as reinforcement from the previous study period. Diet requirements include at least 5 days of food logs each week. Exercise requirements include objective verification of up to 5 exercise sessions per week (as prescribed).
  Interventions: Behavioral: Lifestyle intervention
- Routine care group (No Intervention): Participants in the Routine Care (RC) control group will receive no additional intervention beyond standard of care.

INTERVENTIONS:
Behavioral: Lifestyle intervention — 1. To establish an effective contingency management behavioral program (LIFE), increasing adherence to nutritional recommendations and exercise guidelines during pregnancy.
  2. To examine the impact of the LIFE program on weight gain restriction during pregnancy and postpartum weight loss in obese women in comparison to the RC group.
  3. To examine the impact of the LIFE program on short- and long-term maternal and offspring outcomes at study enrollment, 34-36 weeks gestation and 3 months postpartum in obese women in comparison to the RC group.
  Arms: Lifestyle intervention group

SUMMARY:
Gaining too much weight in pregnancy is associated with adverse pregnancy complications and can have a long-term impact on maternal and offspring health, including increased risk for obesity and metabolic disease. Preventing excessive gestational weight gain could reduce adverse pregnancy outcomes and improve long-term health of mothers and offspring. Thirty obese (BMI ≥30) pregnant women will be recruited for this pilot study and randomly assigned to the Lifestyle Intervention ForEver (LIFE) program or routine care (RC). Participants will be enrolled before 18 weeks gestation and will be followed until 12 weeks after delivery. Women in the LIFE program will be given guidance on healthy eating and exercise at their regularly scheduled obstetric visits. To increase adherence to the program, a contingency management (CM) intervention offering incentives will be used to establish and maintain healthy nutrition and physical activity habits, working towards the goal of restricted weight gain (± 10lb) during their pregnancy. Three study testing visits will be scheduled for all participants: at study entry, 34-36 weeks gestation, and 12 weeks after delivering. Primary outcomes include adherence to the LIFE program, weight change in pregnancy and postpartum, and objective measures of maternal and offspring health.

DETAILED DESCRIPTION:
The ultimate goal of this research is to examine the impact of a healthy lifestyle intervention, targeting weight gain restriction during pregnancy in obese women (BMI≥30kg/m2), on maternal and fetal outcomes.

The overarching research program has 3 main objectives:

1. To establish an effective contingency management behavioral program (LIFE), increasing adherence to nutritional recommendations and exercise guidelines during pregnancy.
2. To examine the impact of the LIFE program on weight gain restriction during pregnancy and postpartum weight loss in obese women in comparison to the RC group.
3. To examine the impact of the LIFE program on short- and long-term maternal and offspring outcomes at study enrollment, 34-36 weeks gestation and 3 months postpartum in obese women in comparison to the RC group.

   * Maternal Outcomes: body composition; peak aerobic capacity; maternal hormonal/metabolic profiles (fasted blood sample); obstetric parameters (incidence of GDM, preeclampsia, cesarean deliveries, obstetric trauma and neonatal complications)
   * Offspring Outcomes: fetal growth pattern (fetal ultrasound); neonatal anthropometry assessed ≤ 48 h of birth (crown-heel length, weight, head, chest and waist circumferences, skinfold analyses); metabolic markers at birth (cord blood); and infant anthropometry at 12 weeks of age (as above).

The experimental hypotheses to be tested are that participation in the LIFE intervention in obese pregnant women will prevent excessive weight gain and/or achieve weight maintenance (± 10 lb) during pregnancy and will result in 7-10% weight loss at 12 weeks postpartum. Secondly, we hypothesize that participation in the LIFE intervention in obese pregnant women will be associated with improved aerobic capacity, reduced incidence of obstetric complications and reduced rates of LGA as a result of beneficial alterations to metabolic intrauterine environment for fetal growth.

With regard to this IRB application, we will be conducting a pilot and feasibility trial to address the following specific aims:

1. To establish the feasibility of the LIFE program as a large-scale funded project, including participant engagement in the intervention and all study visits.
2. To evaluate the feasibility of the LIFE program in achieving weight maintenance and postpartum weight loss targets in obese pregnant women across all three obesity classes.
3. To develop and refine the study materials for the LIFE program and assessment battery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years with a confirmed singleton pregnancy of up to 18 weeks gestation
* Pre-pregnancy or early pregnancy BMI greater than or equal to 30 kg/m2

Exclusion Criteria:

* Aged < 18 years or > 40 years
* BMI < 30 kg/m2 at study screening
* Multiple gestations
* Previously diagnosed with type 1 or type 2 diabetes mellitus
* Subjects will be excluded from the study if they present with any absolute or relative contraindications to exercise in pregnancy (as defined by ACOG); determined by completion of medical questionnaire by supervising physician
* Any evidence of:

  i. Drug or alcohol abuse ii. Presence of any unstable psychiatric disorder iii. Plans to move away from the geographical area within the next nine months iv. Other medical or behavioral factors that, in the judgement of the supervising physician, may interfere with their ability to take part in a lifestyle intervention program during pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measurement of Gestational weight gain from study entry to delivery | Approx. 20-25 weeks
  Maternal weight (lb) will be measured at program entry and at the time of delivery to determine weight gain during the study period.
  Pre-pregnancy body weight will be self-reported and used to estimate total gestational weight gain (lb).

SECONDARY OUTCOMES:
Measure Change from baseline in maternal body composition | 16-21 weeks
  Changes in lean and fat mass will be examined at study entry, in late pregnancy (34-36 weeks gestation) and at 12 weeks postpartum
Measure Change from baseline in maternal aerobic capacity | 16-21 weeks
  Peak aerobic capacity will be examined via a standard maximal oxygen consumption (VO2max) test performed on a stationary cycle ergometer at study entry, in late pregnancy (34-36 weeks gestation), and at 12 weeks postpartum
Measure Maternal hormonal/metabolic changes from baseline | 16-21 weeks
  A fasted blood sample will be collected at study entry, in late pregnancy (34-36 weeks gestation) and at 12 weeks postpartum to examine changes in lipid profile and adipokines (TNF-alpha, leptin). Fasting glucose, insulin and C-peptide will also be measured and entered into the homeostatic model (HOMA) to estimate changes in insulin sensitivity and beta cell function during the study period.
Number of participants with Obstetric complications | 1-25 weeks
  Parameters examined will include:
  * incidence rates of pregnancy complications (gestational diabetes mellitus, preeclampsia, gestational hypertension)
  * examination of obstetric parameters (mode of delivery, incidence of obstetric trauma, neonatal complications)
Change from baseline in maternal dietary intake | 16-21 weeks
  Dietary intake will be examined at study entry (15-18 weeks gestation), in late pregnancy (34-36 weeks gestation) and at 12 weeks postpartum.
Measure Change from baseline in maternal psychometric outcomes | 16-21 weeks
  Psychometric outcomes examined at study entry, in late pregnancy (34-36 weeks gestation) and at 12 weeks postpartum include:
  * Quality of life
  * Depression and mood
  * Physical activity social support
  * Exercise self-efficacy
Measure Offspring - fetal growth | 10-25 weeks
  Fetal growth and abdominal circumference will be examined by fetal ultrasound at approximately 28-30, 34-36 and 38-40 weeks gestation and/or as part of routine care after 28 weeks gestation.
Measure Neonatal size at birth | Within 48 hours of birth
  Between group comparisons of birth size will include birth weight (g), crown-heel length (mm), head circumference (mm), body mass index (kg/m2), ponderal index. Population-specific standard deviation (SD) scores will be calculated and the incidence of small for gestational age, appropriate for gestational age and large for gestational age will be compared between groups.
Measure Neonatal body composition at birth | Within 48 hours of birth
  Neonatal lean and fat mass (g) will be calculated based on anthropometric measurements performed within 48 hours after birth
Measure Offspring metabolic markers | 20-25 weeks
  Concentrations of insulin-like growth factor (IGF)-I, IGF-II, IGF binding protein-1, IGF binding protein-3, glucose, insulin, leptin and triglyceride will be examined from cord blood samples taken at the time of delivery.
Measure Pilot study outcomes | 32-37 weeks
  The following pilot and feasibility outcomes will be assessed:
  * Participant recruitment rate (number of participants recruited per week)
  * Participant retention rate (percentage of participants completing all outcomes)
  * Adherence to the study program (completion of study data, food records, exercise sessions)
  * Success of the study program (percentage of participants achieving target gestational weight gain of plus/minus 10 lb)
  * Intervention dose (total intervention time in hours).
Measure Postpartum weight retention at 12 weeks postpartum | 12 weeks
  Maternal weight (lb) will be measured at 6 & 12 weeks postpartum and compared to delivery weight (lb) to determine postpartum weight retention.
Measure Change from baseline in maternal physical activity levels | 16-21 weeks
  Physical activity levels will be examined at study entry (15-18 weeks gestation), in late pregnancy (34-36 weeks gestation) and at 12 weeks postpartum.
Measure Infant size at 12 weeks of age | 12 weeks
  Between group comparisons of body weight (g), length (mm), head circumference (mm), body mass index (kg/m2), and ponderal index. Population-specific SD scores will be calculated and compared between groups.
Measure Infant body composition at 12 weeks of age | 12 weeks
  Infant lean and fat mass (g) will be calculated based on anthropometric measurements performed at 12 weeks of age.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Catanzaro, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States